CLINICAL TRIAL: NCT00786695
Title: Esomeprazole as a Diagnostic Test for Gastroesophageal Reflux Disease in Patients With Noncardiac Chest Pain
Brief Title: Study Using Esomeprazole as a Diagnostic Test for GERD in Patients With NCCP
Acronym: ECP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Khek Yu Ho / Professor, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: D/00/764
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: noncardiac chest pain; gastroesophageal reflux disease; diagnostic test; proton pump inhibitor; esomeprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Identical looking Placebo
  Interventions: Drug: Placebo
- esomeprazole (Experimental): esomeprazole (40 mg o d) for 14 days
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — esomeprazole (40 mg o d) for 14 days
  Other Names: nexium
  Arms: esomeprazole
Drug: Placebo — Identical looking Placebo, same regimen, for 14 days
  Arms: Placebo

SUMMARY:
Gastroesophageal reflux disease (GERD), with its cardinal symptom, heartburn, is the most common disorder of the esophagus in the West. Comparatively, GERD is less common in Singapore but its frequency in the population is increasing. Although the vast majority of patients with GERD have heartburn and acid regurgitation, GERD can present in atypical ways, including as a non-cardiac chest pain (NCCP). We have previously shown that GERD is a common cause of NCCP in Singapore. Up to 40% of our patients with NCCP had endoscopic esophagitis, abnormal 24-hour pH monitoring results, and/or a positive acid perfusion test. These tests, although diagnostic, are costly, labour intensive, and not always readily available in the primary care setting. A trial of high-dose proton pump inhibitor (e.g. omeprazole 60 mg daily) has been proposed as a simple, safe, non-invasive and reliable means to diagnose GERD in Western patients with NCCP. We have not used the test routinely in our practice. This study will evaluate the use of a short course of esomeprazole, the S-isomer of omeprazole, as a diagnostic test for detecting GERD in patients with NCCP. The hypothesis is that in NCCP patients with GERD, esomeprazole will resolve their symptoms. Consecutive patients diagnosed with NCCP at the National University Hospital, Singapore, will be invited to participate in the study. Eligible patients will be randomly assigned to receive either esomeprazole (40 mg o d) for 14 days, or comparable dose of placebo at a similar schedule for 14 days, in a double-blinded fashion. At the start of the study, all subjects will complete a baseline symptom assessment. Symptoms will be scored on a graded scale based on severity. During the study weeks, each patient will record his/her own daily symptoms. The patient will be assessed again after the 14-day treatment. The primary outcome measure will be the change in symptom score after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent chest pain of more than three months duration with either (1) normal or non-obstructive coronary arteries (<50% luminal diameter narrowing), (2) normal dobutamine stress echocardiography or (3) a negative exercise electrocardiogram and a cardiologist's evaluation that symptoms are not cardiac in origin.

Exclusion Criteria:

* Patients will be excluded if they are < 18 or > 70 years old, are pregnant, have a medical contraindication for esomeprazole therapy, have already been empirically treated with an antireflux regimen, report a history of peptic ulcer disease or gastrointestinal surgery, or are unwilling or unable to provide informed consent. In addition, patients who are unable to fully complete all stages of the study will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
symptom resolution | 14 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Ho KY. Gastroesophageal reflux disease is uncommon in Asia: evidence and possible explanations. World J Gastroenterol. 1999 Feb;5(1):4-6. doi: 10.3748/wjg.v5.i1.4. No abstract available. PMID 11819371
- [Background] Lim LG, Ho KY. Gastroesophageal reflux disease at the turn of millennium. World J Gastroenterol. 2003 Oct;9(10):2135-6. doi: 10.3748/wjg.v9.i10.2135. PMID 14562363
- [Background] Ho KY. Gastroesophageal reflux disease in Asia: a condition in evolution. J Gastroenterol Hepatol. 2008 May;23(5):716-22. doi: 10.1111/j.1440-1746.2008.05380.x. PMID 18410606
- [Background] Ho KY, Gwee KA, Khor JL, Selamat DS, Yeoh KG. Validation of a graded response questionnaire for the diagnosis of gastroesophageal reflux disease in an Asian primary care population. J Clin Gastroenterol. 2008 Jul;42(6):680-6. doi: 10.1097/MCG.0b013e3180653613. PMID 18347510
- [Background] Ho KY, Cheung TK, Wong BC. Gastroesophageal reflux disease in Asian countries: disorder of nature or nurture? J Gastroenterol Hepatol. 2006 Sep;21(9):1362-5. doi: 10.1111/j.1440-1746.2006.04341.x. PMID 16911677
- [Background] Lim SL, Goh WT, Lee JM, Ng TP, Ho KY; Community Medicine GI Study Group. Changing prevalence of gastroesophageal reflux with changing time: longitudinal study in an Asian population. J Gastroenterol Hepatol. 2005 Jul;20(7):995-1001. doi: 10.1111/j.1440-1746.2005.03887.x. PMID 15955205
- [Background] Ho KY, Kang JY, Yeo B, Ng WL. Non-cardiac, non-oesophageal chest pain: the relevance of psychological factors. Gut. 1998 Jul;43(1):105-10. doi: 10.1136/gut.43.1.105. PMID 9771413
- [Background] Ho KY, Kang JY, Seow A. Prevalence of gastrointestinal symptoms in a multiracial Asian population, with particular reference to reflux-type symptoms. Am J Gastroenterol. 1998 Oct;93(10):1816-22. doi: 10.1111/j.1572-0241.1998.00526.x. PMID 9772037
- [Background] Ho KY, Kang JY, Seow A. Patterns of consultation and treatment for heartburn: findings from a Singaporean community survey. Aliment Pharmacol Ther. 1999 Aug;13(8):1029-33. doi: 10.1046/j.1365-2036.1999.00571.x. PMID 10468677
- [Background] Ho KY, Kang JY. Reflux esophagitis patients in Singapore have motor and acid exposure abnormalities similar to patients in the Western hemisphere. Am J Gastroenterol. 1999 May;94(5):1186-91. doi: 10.1111/j.1572-0241.1999.01063.x. PMID 10235190